CLINICAL TRIAL: NCT05722288
Title: A Randomized, Phase II Clinical Trial of Time-Restricted Eating Versus Nutritional Counseling in Cancer Patients Receiving Radiation or Chemoradiation to Evaluate Its Impact on Toxicity and Efficacy
Brief Title: Time-Restricted Eating Versus Nutritional Counseling for the Reduction of Radiation or Chemoradiation Tx Side Effects in Patients With Prostate, Cervical, or Rectal Cancers
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 21709; NCI-2023-00238 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21709 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2023-01-23; First posted 2023-02-10 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Localized Prostate Carcinoma; Locally Advanced Cervical Carcinoma; Locally Advanced Rectal Carcinoma; Malignant Solid Neoplasm; Recurrent Prostate Carcinoma; Stage I Prostate Cancer AJCC v8; Stage IB Cervical Cancer FIGO 2018; Stage IB2 Cervical Cancer FIGO 2018; Stage II Prostate Cancer AJCC v8; Stage II Rectal Cancer AJCC v8; Stage IIA Cervical Cancer FIGO 2018; Stage IIB Cervical Cancer FIGO 2018; Stage III Prostate Cancer AJCC v8; Stage III Rectal Cancer AJCC v8; Stage IIIA Cervical Cancer FIGO 2018; Stage IIIB Cervical Cancer FIGO 2018; Stage IIIC Cervical Cancer FIGO 2018; Stage IVA Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms; Rectal Neoplasms | interventions — Specimen Handling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm I (time-restricted eating) (Experimental): Patients undergo time-restricted eating Monday through Friday only of each week on study during standard RT or chemoRT. Patients also undergo collection of blood throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Behavioral: Short-Term Fasting
- Arm II (nutritional counseling) (Active Comparator): Patients receive nutritional counseling on study. Patients also undergo collection of blood throughout the trial.
  Interventions: Procedure: Biospecimen Collection; Other: Informational Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Other: Informational Intervention — Receive nutritional counseling
  Arms: Arm II (nutritional counseling)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Behavioral: Short-Term Fasting — Undergo time-restricted eating
  Other Names: Intermittent Fasting; Short-term Intermittent Fasting
  Arms: Arm I (time-restricted eating)

SUMMARY:
This phase II trial studies how well time-restricted eating works in reducing side effects of radiation or chemoradiation side effects when compared to nutritional counseling among patients with prostate, cervical, and rectal cancers. Time-restricted eating, also called short term fasting or intermittent fasting, is an eating plan that alternates between not eating food (fasting) and non-fasting periods. Nutritional counseling involves being asked to follow a healthy, balanced diet that includes instructions on what kinds of food are better tolerated during radiation and chemoradiation therapy. This trial may help researchers determine if certain diets may improve the anti-cancer effects of radiation therapy and reduce the side-effects of this treatment. If successful, these diets may be integrated into the future treatment of prostate, cervical, and rectal cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To test the hypothesis that time-restricted eating during radiation therapy (RT) or chemotherapy and radiation therapy (chemoRT) could reduce the level of accumulated double stranded deoxyribonucleic acid (dsDNA) damage in peripheral blood mononuclear cells (PBMCs) over the course of RT as measured by the gH2ax assay.

II. To examine if time-restricted eating during RT is associated with reduced toxicity as measured by clinician reported adverse events using Common Terminology Criteria for Adverse Events (CTCAE) version (v)5.0, improved patient quality of life as measured by European Organization for the Research and Treatment of Cancer Quality of Life (EORTC-PR25) (prostate cancer) and EORTC-CR29 (rectal cancer), reduced dsDNA damage as measured by assay for 8-oxo-dG and persistent DNA damage in shed epithelial cells from the urinary tract, reduced oxidative DNA damage as measured by reduced cumulative 8-oxoguanine DNA adducts, impacts the diversity of microbiome in relation and development of radiation induced microbiota dysbiosis and metabolic impact using liquid chromatography mass spectrometry (LC/MS) metabolomic analysis and correlative serological markers including IGF-1.0).

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients undergo time-restricted eating Monday through Friday only of each week on study during standard RT or chemoRT. Patients also undergo collection of blood throughout the trial.

ARM II: Patients receive nutritional counseling on study. Patients also undergo collection of blood throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 or older
* Localized high risk prostate cancer or node positive prostate cancer histologically confirmed by biopsy or recurrence after surgical resection planning to receive whole pelvis radiation therapy +/- androgen deprivation therapy or
* Locally advanced cervical cancer receiving whole pelvic/paraaortic radiation therapy + concurrent cisplatin-based chemotherapy or
* Locally advanced rectal cancer receiving whole pelvis radiation therapy + concurrent 5FU/capecitabine
* Eastern Cooperative Oncology Group (ECOG) Performance Status 0-2
* Able to provide a written consent for study participation

Exclusion Criteria:

* PROSTATE CANCER: Prior radiation therapy to the prostate gland or pelvis
* PROSTATE CANCER: Prior therapy with androgen deprivation therapy for longer than 6 months
* PROSTATE CANCER: Prior chemotherapy
* PROSTATE CANCER: Men with diabetes may enroll, provided they are on stable doses of antihyperglycemic medication for at least 6 months and provided the physician managing their diabetes feels they can safely hold antihyperglycemic medication during daily time-restricted eating
* PROSTATE CANCER: Must be eligible to receive neoadjuvant and concurrent androgen deprivation therapy, but androgen deprivation therapy is not required
* PROSTATE CANCER: Men whose treatment plan includes up-front docetaxel will be excluded due potential confounding
* PROSTATE CANCER: Patients whose body mass index (BMI) is less than 21 at time of screening
* PROSTATE CANCER: Men who are currently undergoing a strict macronutrient or time limited diet including ketogenic, low-carbohydrate (carb), paleolithic (paleo), or warrior diet are excluded
* GYNECOLOGIC CANCER: Prior radiation therapy to the cervix, uterus or pelvis
* GYNECOLOGIC CANCER: Prior chemotherapy
* GYNECOLOGIC CANCER: Women must not be pregnant, planning to become pregnant or lactating at the time of enrollment or during the course of the study
* GYNECOLOGIC CANCER: Women with diabetes may enroll, provided they are on stable doses of antihyperglycemic medication for at least 6 months and provided the physician managing their diabetes feels they can safely hold antihyperglycemic medication during daily time-restricted eating
* GYNECOLOGIC CANCER: Must be eligible to receive chemotherapy that is cisplatin based
* GYNECOLOGIC CANCER: Patients whose BMI is less than 21 at time of screening
* GYNECOLOGIC CANCER: Women who are currently undergoing a strict macronutrient or time limited diet including ketogenic, low-carb, paleo, or warrior diet are excluded
* RECTAL CANCER: Prior pelvic radiation therapy
* RECTAL CANCER: Prior chemotherapy
* RECTAL CANCER: Patients with diabetes may enroll, provided they are on stable doses of antihyperglycemic medication for at least 6 months and provided the physician managing their diabetes feels they can safely hold antihyperglycemic medication during daily time-restricted eating
* RECTAL CANCER: Patients whose BMI is less than 21at time of screening
* RECTAL CANCER: Women must not be pregnant, planning to become pregnant or lactating at the time of enrollment or during the course of the study
* RECTAL CANCER: Patients who are currently undergoing a strict macronutrient or time limited diet including ketogenic, low-carb, paleo, or warrior diet are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2026-07-20 (Estimated); Study Completion 2026-07-20 (Estimated)

PRIMARY OUTCOMES:
Cumulative double strand deoxyribonucleic acid (dsDNA) damage of normal tissue | Up to 1 year after radiation therapy/chemotherapy and radiation therapy (chemoRT)
  Will be measured by the gH2ax assay. The study population will be described by, and randomized groups compared with respect to baseline characteristics including demographics (age, race/ethnicity, education, gender for rectal cancer), clinical characteristics (prostate: pre-treatment prostate-specific antigen [PSA], National Comprehensive Cancer Network [NCCN] staging and rectal: American Joint Committee on Cancer version 8 [AJCC8] staging), and metabolic features (diabetes, HbA1c, waist circumference, fat mass, lipids). Given the potential for differential outcomes among diabetics, the analysis of trial outcomes will also include diabetes as a covariate.
Percentage of patients completing 4 weeks of time-restricted eating during RT | Up to 4 weeks
  Feasibility and tolerability is pre-determined to be met if least 70% of patients randomized to time-restricted eating can complete at 4 weeks of time-restricted eating during their radiation course. Will be assessed through quarterly assessments of missing data points. The study dietician will track and report on compliance in the intervention (time-restricted eating) arm, and research coordinator will track and report accrual, screen failures, self-reporting survey completions and data entry metrics. Trouble areas will be discussed, and protocol amendments developed accordingly. The co-principal investigators (PIs) will review and determine whether feasibility of analysis is impacted and whether corrective measures can be implemented to improve data completeness.

SECONDARY OUTCOMES:
Rates of objective clinical adverse events (AEs) | Up to 6 months
  Will assess acute (during and at 4 weeks after treatment) and long term (at 3 or 6 months). Will use repeated measures analysis of variance (ANOVA) accounting for within-between interactions. Will also perform simple paired t-tests to evaluated differences in toxicity observed by clinicians at the two final post-RT time points to evaluate if there is a trend towards clinical benefit associated with fasting.
Quality of life (QoL) indices - PR25 | Up to 1 year after completion of RT/chemoRT
  Will be measured by previously validated instruments for QoL studies in prostate and rectal cancer patients, European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire - Prostate (EORTC-QLQ-PR25) during and after treatment. AEs will be clinician collected during study visits while QoL surveys will be collected from patients directly through automated electronic surveys. Will use repeated measures ANOVA accounting for within-between interactions.
Quality of life (QoL) indices - CR29 | Up to 1 year after completion of RT/chemoRT
  Will be measured by previously validated instruments for QoL studies in prostate and rectal cancer patients, European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire - Prostate EORTC-QLQ-Colorectal (CR29) during and after treatment. AEs will be clinician collected during study visits while QoL surveys will be collected from patients directly through automated electronic surveys. Will use repeated measures ANOVA accounting for within-between interactions.
Accumulated gH2ax foci | Up to 1 year after completion of RT/chemoRT
  Will represent persistent damage in shed epithelial cells from the urinary tract and peripheral blood mononuclear cells (PBMCs) by flow cytometry. Will use repeated measures ANOVA accounting for within-between interactions.
Oxidative DNA damage | Up to 1 year after completion of RT/chemoRT
  Will be measured by reduced cumulative 8-oxoguanine DNA adducts. Will use repeated measures ANOVA accounting for within-between interactions.

CONTACTS AND LOCATIONS:
Overall Officials: Yun R Li, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States